CLINICAL TRIAL: NCT03199716
Title: Parent Mentors to Improve Adherence to Type I Diabetes Care Regimen in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 615897
Record Dates: First submitted 2015-02-19; First posted 2017-06-27 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent Mentors and Intervention Group (Experimental): Parent mentors are parents from our UC Davis Pediatrics Endocrinology clinic who have met our parent mentor inclusion criteria; the intervention group are families in our clinic who have met our mentee family inclusion criteria
  Interventions: Other: Parent mentors
- Control Group with no Parent Mentors (No Intervention): The control group is made up of families at our UC Davis Pediatrics Endocrinology clinic who have met the mentee family inclusion criteria but are not matched with a parent mentor

INTERVENTIONS:
Other: Parent mentors — Parent mentors are to meet up with their assigned intervention group 4 times in 1 year and call the families monthly to document any diabetic complications
  Arms: Parent Mentors and Intervention Group

SUMMARY:
The study aim is to determine if parent mentors can improve adherence to the intensive multiple daily injection regimen (MDI) or the insulin pump therapy, through monitoring the frequency of blood glucose measurements. Researchers are also trying to determine if the parent mentors can improve glycemic control, which is measured through HbA1c. The study hypothesis is that trained parent mentors can help families with children who have poorly controlled T1DM improve adherence to their diabetes regimen and improve their metabolic control.

DETAILED DESCRIPTION:
The study aim is to determine if parent mentors can improve adherence to the intensive multiple daily injection regimen (MDI) or the insulin pump therapy, through monitoring the frequency of blood glucose measurements. Researchers are also trying to determine if the parent mentors can improve glycemic control, which is measured through HbA1c. Diabetic knowledge, responsibility for diabetes care, degree of diabetes related family conflicts, and major complications of diabetes will also be collected during the patient's routine clinic visit. The study hypothesis is that trained parent mentors can help families with children who have poorly controlled T1DM improve adherence to their diabetes regimen and improve their metabolic control.

ELIGIBILITY:
Inclusion Criteria for mentee families:

* Residing within 60 miles of a Parent Mentor
* Child diagnosed with T1DM greater than or equal to 1 year at the start of our study's data collection (February 2015)
* On multiple daily injection regime or insulin pump therapy
* Mean HbA1c between 8.5 - 12.5% over the last 2 clinic visits

Inclusion Criteria for parent mentors:

* Child diagnosed with T1DM greater than or equal to 2 years at the start of our study's data collection
* Compliant with suggestions made by the diabetes care team
* Mean HbA1c less than or equal to 8% over the last 2 clinic visits
* No episodes of diabetic ketoacidosis, aside from initial episode at diagnosis, if applicable

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-03-23 (Actual); Study Completion 2017-03-23 (Actual)

PRIMARY OUTCOMES:
Daily frequency of blood glucose monitoring (BGM) | up to 12 months
  Number of glucose monitoring events per day

SECONDARY OUTCOMES:
HbA1c levels | up to 12 months
  Values of HbA1c in blood

OTHER OUTCOMES:
Diabetes knowledge | up to 12 months
  Score measured by Diabetes Numeracy Test (DNT-15)
Degree of diabetes related family conflicts | up to 12 months
  Score based on Questionnaire (r-DFCS)
Responsibility for diabetes care | up to 12 months
  Score based on Diabetes Family Responsibility Questionnaire (DFRQ)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Styne, MD, Principal Investigator — UC Davis Pediatrics Endocrinology; Yvonne Lee, MD, Principal Investigator — UC Davis Pediatrics Endocrinology
Locations (1):
- UC Davis Pediatrics Endocrinology, Sacramento, California, United States